CLINICAL TRIAL: NCT05089396
Title: Assessment of Dentoskeletal Effects Concomitant With Skeletally Anchored Maxillary Protraction in Orthodontic Skeletal Class III Patients
Brief Title: Effects of Conventional Versus Skeletally Anchored Facemask in Treatment of the Prepubertal Skeletal Class III Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Amr Mohamed Gouda Embaby, Dentist, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SA maxillary protraction
Record Dates: First submitted 2021-10-11; First posted 2021-10-22 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Maxillary Deficiency; Maxillary Retrusion
MeSH Terms: conditions — Retrognathia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional dentally anchored maxillary protraction (Active Comparator): A petit facemask will be used for maxillary protraction along with a facemask splint (two acrylic bite blocks connected through a transpalatal arch). a force of 380 gm to 400 gm will be applied through the extra-oral elastics the will be attached to the facemask on one side and to the facemask splint on the other side.
  Interventions: Other: Maxillary protraction
- skeletally anchored maxillary protraction (Experimental): A petit facemask will be used for maxillary protraction along with a facemask splint (two acrylic bite blocks connected through a transpalatal arch) in addition, two miniscrews will be inserted in the anterior region of the palate one on each side of the midline to provide skeletal anchorage for the facemask splint. a force of 380 gm to 400 gm will be applied through the extra-oral elastics the will be attached to the facemask on one side and to the facemask splint on the other side.
  Interventions: Other: Maxillary protraction

INTERVENTIONS:
Other: Maxillary protraction — A petit facemask will be used for maxillary protraction along with a facemask splint (two acrylic bite blocks connected through a transpalatal arch) in the active comparator group. in the experimental group, two miniscrews will be inserted in the anterior region of the palate one on each side of the midline to provide skeletal anchorage for the facemask splint. in both groups, a force of 380 gm to 400 gm will be applied through the extra-oral elastics the will be attached to the facemask on one side and to the facemask splint on the other side.

SUMMARY:
The aim of this study will be directed to the assessment of dentoskeletal effects concomitant with skeletally anchored maxillary protraction in orthodontic skeletal Class III patients.

DETAILED DESCRIPTION:
Skeletal Class III is a challenging problem that is confronting orthodontists in their everyday orthodontic practice. The prevalence of this malocclusion varies globally among and within populations with the greatest incidence among Asian countries. It was reported that Class III malocclusion represents 3.98% and 5.93% of malocclusions in mixed and permanent dentitions respectively. Among Egyptians, the prevalence of Class III malocclusion during mixed dentition was found to be 5.9 % according to the sample studied by Fsifis et al.

Different skeletal components contribute to the development of the classic Class III with convex or straight profiles. These components are either maxillary retrognathism, mandibular prognathism relative to other craniofacial structures, or even a combination of them. According to the sample studied by Ellis and Macnamara, they found 65% to 67% of skeletal Class III was due to maxillary skeletal retrusion.

The growth and severity of the sagittal skeletal discrepancy dictate the possible treatment modalities. On one hand, Growth modification is indicated in individuals who have not reached the growth spurt yet. On the other hand, cessation of growth leaves only orthodontic camouflage and orthognathic surgery as treatment options, the severity of the anteroposterior discrepancy and dental compensation determine which of them gives the best clinical results.

The most common approach for the treatment of growing Class III patients with maxillary retrognathism is the facemask (FM) accompanied by rapid maxillary expansion (RME). RME was claimed to open the midpalatal suture and affect the other nine sutures adjacent to the maxilla. Accordingly, it is said to facilitate the orthopedic effect of the facemask. However, a meta-analysis concluded that treatment with facemask with or without RME is clinically effective with a nonsignificant difference.

Forces from protraction facemask are applied to dental structures so, it has side effects as mesial movement and extrusion of maxillary molars, proclination of upper incisors, retroclination of mandibular incisors, backward rotation of the mandible, and increase in the lower facial height. These side effects might be desirable or undesirable according to the clinical situation.

Maximizing skeletal effects and minimizing dental effects will reduce the tendency for relapse and might be a desirable clinical outcome. For this purpose, in 1985 Kokich et al used ankylosed canines as a form of absolute anchorage for maxillary protraction. The advent of temporary anchorage devices (TADs) led to many reports with skeletally anchored maxillary protraction, Singer et al, Enacar et al, Hong et al, and Kircelli et al.

This was followed by several studies applying facemask to miniplates at the zygomatic buttress, lateral nasal wall, and miniscrews (MS) in the zygomatic buttress, or in the palate. Consequently, the present study will be directed to evaluate the effects of skeletally anchored maxillary protraction.

ELIGIBILITY:
Inclusion Criteria:

* Growing Class III patients with a prepubertal stage of skeletal maturity according to the cervical vertebral maturation method.
* Skeletal Class III malocclusion with maxillary deficiency (ANB, <0°; N perp-A<1mm) with or without mild mandibular prognathism.
* Late mixed or early permanent dentition at the start of treatment characterized by a Wits appraisal of -1 mm or less and an Angle Class III molar relationship or anterior crossbite.
* Vertically normal growth pattern determined by cephalometric radiographs.
* Patients are free from developmental or congenital conditions such as cleft lip/palate or other craniofacial anomalies.
* No previous orthodontic treatment.

Exclusion Criteria:

* Poor oral hygiene or periodontally compromised patient.
* Patients with craniofacial anomalies or previous history of trauma, bruxism, or parafunctions.
* Previous orthodontic treatment.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 14 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
midfacial length | 1 year
  linear distance between condylon and A points

CONTACTS AND LOCATIONS:
Locations (1):
- Al-azhar university- Faculty of Dental Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seiryu M, Ida H, Mayama A, Sasaki S, Sasaki S, Deguchi T, Takano-Yamamoto T. A comparative assessment of orthodontic treatment outcomes of mild skeletal Class III malocclusion between facemask and facemask in combination with a miniscrew for anchorage in growing patients: A single-center, prospective randomized controlled trial. Angle Orthod. 2020 Jan;90(1):3-12. doi: 10.2319/101718-750.1. Epub 2019 Aug 12. PMID 31398066